CLINICAL TRIAL: NCT00767793
Title: A Multi-Center, Double-Masked, Randomized, Placebo-Controlled, Ascending Dose Study of INS117548 Ophthalmic Solution in Subjects With Bilateral Ocular Hypertension or Early Primary Open Angle Glaucoma
Brief Title: A Placebo-Controlled Study of INS117548 Ophthalmic Solution in Subjects With Glaucoma (P08650)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P08650; 037-101
Record Dates: First submitted 2008-10-02; First posted 2008-10-07 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Arm 1 (Placebo Comparator): One drop in each eye every 12 hours for seven days
  Interventions: Drug: Placebo
- Arm 2 (Experimental): One drop of Concentration #1 in one eye and one drop of placebo in contralateral eye every 12 hours for seven days
  Interventions: Drug: INS117548
- Arm 3 (Experimental): One drop of Concentration #2 in one eye and one drop of placebo in contralateral eye every 12 hours for seven days
  Interventions: Drug: INS117548
- Arm 4 (Experimental): One drop of Concentration #3 in one eye and one drop of placebo in contralateral eye every 12 hours for seven days
  Interventions: Drug: INS117548

INTERVENTIONS:
Drug: Placebo — One drop in each eye every 12 hours for seven days
  Arms: Arm 1
Drug: INS117548 — One drop of Concentration #1 in one eye and one drop of placebo in contralateral eye every 12 hours for seven days
  Arms: Arm 2
Drug: INS117548 — One drop of Concentration #2 in one eye and one drop of placebo in contralateral eye every 12 hours for seven days
  Arms: Arm 3
Drug: INS117548 — One drop of Concentration #3 in one eye and one drop of placebo in contralateral eye every 12 hours for seven days
  Arms: Arm 4

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of INS117548 ophthalmic solution.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of bilateral ocular hypertension or early primary open angle glaucoma
* Have best corrected visual acuity in both eyes of at least +0.5 or better

Exclusion Criteria:

* Are diagnosed with closed angle glaucoma, exfoliation syndrome or exfoliation glaucoma, and pigment dispersion or secondary glaucoma
* Have a history of any type of intraocular surgery, except for cataract surgery
* Have had cataract surgery within three months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 15
Rate of discontinuation | 15
Changes in: >Ophthalmic exam parameters >Corneal thickness >Intraocular pressure >Visual Acuity >Physical exam, vital signs and laboratory parameters | 15
Compliance | 15

CONTACTS AND LOCATIONS:
Overall Officials: Reza Haque, MD, PhD, Study Director — Medical Monitor, Inspire